CLINICAL TRIAL: NCT07342439
Title: Phase 3 Study of Serine Supplementation to Protect Vision in MacTel
Brief Title: Study of Serine Supplementation to Protect Vision in MacTel
Acronym: SEErine
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Lowy Medical Research Institute Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2026-001
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Macular Telangiectasia Type 2 (MacTel)
Keywords: Serine; MacTel
MeSH Terms: interventions — Serine

STUDY DESIGN:
Intervention Model Description: masked, two-arm, parallel-group, randomized, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- L-serine (Experimental): Participant receives oral L-serine
  Interventions: Drug: L-serine
- Placebo (Placebo Comparator): Participant receives placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: L-serine — L-serine powder administered twice daily
  Arms: L-serine
Other: Placebo — Placebo powder administered twice daily
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to look at the efficacy and safety of giving oral serine (an amino acid) on the progression of structural and functional changes of the retina in people with MacTel type 2. The main questions it aims to answer are:

* Does serine slow the progression of MacTel?
* Is long-term serine supplementation safe in people with MacTel? Researchers will compare serine to a placebo (a look-alike substance that contains no drug) to see if serine works to slow the progression of MacTel.

Participants will:

* Take serine or a placebo twice a day for 24 months
* Visit the clinic once every 6 months for eye exam, eye imaging and blood tests
* Keep a diary of their symptoms, missed doses, and changes in medications

DETAILED DESCRIPTION:
Macular telangiectasia type 2 (MacTel) is a bilateral, slowly progressive retinal neurodegenerative disease characterized by photoreceptor loss, vascular abnormalities, and gradual decline in visual function.

Alterations in serine metabolism and the accumulation of toxic deoxysphingolipids have been implicated in the pathophysiology of MacTel. Oral serine supplementation has been proposed as a potential approach to modify this metabolic pathway and reduce the formation of potentially neurotoxic metabolites.

This study is a randomized, double-masked, placebo-controlled, parallel-group clinical trial designed to evaluate the effect of oral serine supplementation on disease progression in participants with macular telangiectasia type 2.

Participants will undergo a screening evaluation to determine eligibility. Eligible participants will be adults aged 18 years or older with a confirmed diagnosis of MacTel through the Natural History Observation Registry (NHOR) study. Participants must meet all eligibility criteria. Eligibility and assignment of the study eye will be determined by review of the images taken at screening. If both eyes are eligible, both eyes may be included as study eyes. A minimum of 110 participants will complete the study.

At the baseline visit, participants will be randomized in a 1:1 ratio to receive either oral serine or placebo. Randomization will be stratified by diabetes status to ensure balanced distribution of participants with and without type 2 diabetes between treatment groups. Participants, investigators, study staff, and outcome assessors will remain masked to treatment assignment throughout the study.

Participants will receive their assigned study treatment for 24 months. In-person study visits will occur every 6 months, with telephone contacts between visits to assess treatment compliance and adverse events. Retinal structure, visual function, and participant safety will be monitored throughout the 24-month treatment period. A follow-up telephone contact will occur approximately 4 weeks after discontinuation of study treatment.

Data will be collected on both eyes of each participant; however, only eyes designated as study eyes and meeting eligibility criteria will be included in the primary efficacy analysis.

The primary objective of the study is to evaluate the effect of serine supplementation compared with placebo on the progression of photoreceptor loss in MacTel. Secondary objectives include the effect of serine supplementation on further structural retinal changes and visual function as well as the assessment of safety and tolerability of long-term oral serine supplementation in this population.

ELIGIBILITY:
Inclusion Criteria

* Be able to read, comprehend, and agree to conditions as explained in the informed consent document and provide written informed consent;
* Be at least 18 years of age;
* Enrolled or enrolling in the Natural History Observation and Registry Study (NHOR) and confirmed with MacTel type 2 by the Reading Center in at least one eye*;
* Participant has clear ocular media (both eyes) for sufficient image quality;
* Participant must have steady fixation in the foveal or parafoveal area;
* Female participants of childbearing potential must agree to use a highly effective method of contraception from the time consent is signed until six days after treatment discontinuation (this is due to a lack of safety data on use of L-serine in pregnant and breastfeeding women; and to allow for medication wash out post treatment discontinuation). Highly effective methods of contraception include:

  (i)Combined hormonal contraception associated with inhibition of ovulation, (ii) progesterone only hormonal contraception associated with inhibition of ovulation (iii) Intrauterine devices, (iv) surgical sterilization such as bilateral tubal occlusion or vasectomized partner or (v) true abstinence (refraining from heterosexual intercourse during the entire period associated with the study treatments, and the reliability of sexual abstinence is in line with the usual lifestyle of the subject)
* Willing and able to comply with study protocol and follow-up visits
* Agree to unconditional use of their donated samples, images and/or data;
* Be able to fast for at least 10 hours prior to blood specimen collection;
* Have a minimum area of total EZ loss of 0.16 mm2 in the study eye. The Reading Center will determine the exact size once images are uploaded.
* Participant has a BCVA of better than or equal to 20/100 Snellen equivalent (>/= 50 letters) using Early Treatment Diabetic Retinopathy Study (ETDRS) charts at a starting distance of 4 meters in the study eye.

Exclusion Criteria:

* Unable to undergo the study procedures or unavailable for follow up visits;
* Unwilling to agree to blanket consent for use of the acquired data, including human biological specimens and images;
* Participant is pregnant, breastfeeding or planning a pregnancy during the study time period;
* Participant has taken serine or glycine supplements in the last 3 months;
* Participant is currently taking or has been taking Fibrates such as fenofibrate, clofibrate, ciprofibrate, bezafibrate, gemfibrozil within the last 3 months;
* Participant has known allergy or hypersensitivity to serine or rice;
* Participant is currently taking or has been taking tamoxifen, chloroquine (or hydroxychloroquine) and/or other retinotoxic substances; for a total period of 6 months
* Participant has uncontrolled type 1 or type 2 diabetes (defined as an HbA1c level of 9% or higher at screening (with or without medication);
* Participant has uncontrolled hypo- or hyperthyroidism, defined as TSH-levels of below 0.4mU/L or above 4.0mU/L at screening with or without treatment;
* Participant is undergoing chemotherapy, radiation therapy or other treatments for active cancer;
* Participant has significant kidney disease or an estimated glomerular filtration rate <50 ml/min/1.73m2 at screening;
* Participant has an active and/ or chronic liver disease (including viral hepatitis, autoimmune liver disease, hemochromatosis, homozygous alpha1-antitrypsin deficiency and Wilson disease, primary biliary cirrhosis, primary sclerosing cholangitis) or poor liver function as estimated by transaminases (ALT/AST) or gamma glutamyl transferase (GGT) or alkaline phosphatase or bilirubin above 2xULN (upper limit of normal) at screening;
* Participant is currently enrolled in another clinical treatment trial or participated in one within the last 30 days;
* Participant has previously received a CNTF device ("Encelto"; either eye) or has intentions of receiving a CNTF device in either eye during the duration of this study;
* Participant shows signs of retinal diseases other than MacTel (including central serous chorioretinopathy, severe non-proliferative or proliferative diabetic retinopathy, diabetic macular edema, age-related macular degeneration, preretinal membrane) that, in the judgment of the investigator, may confound the diagnosis, procedures or outcome of the study (either eye);
* Participant has a diagnosis of uncontrolled glaucoma with intraocular pressure of >30 mm Hg (despite current pharmacological or non-pharmacological treatment; either eye);
* Participant has evidence of pathologic myopia in either eye;
* Participant has significant corneal or media opacities in either eye;
* Participant has any of the following lens opacities: cortical opacity > standard 3, posterior subcapsular opacity > standard 2, or a nuclear opacity > standard 3 as measured on the Age-Related Eye Disease Study (AREDS) clinical lens grading system (either eye);
* Participant has undergone lens removal in the previous 3 months or YAG laser within the last 4 weeks, in either eye;
* Participant has a chronic requirement (eg, ≥ 4 weeks at a time) for ocular medications (vitamins, supplements and artificial tears are permitted) and/or has a diagnosed disease that, in the judgment of the examining physician, may be vision threatening or may affect the primary outcome in the study eye;
* Participant has had previous ocular treatments that in the judgment of the investigator may complicate the evaluation of the central retina (including vitreo-retinal surgeries, central laser treatments, including central non-damaging retinal laser therapy (either eye); previous peripheral laser treatments or cryotherapy are NOT exclusionary;
* Participant has ever received any periocular or intravitreal injections (including intravitreal anti-vascular endothelial growth factor (anti-VEGF), periocular or intravitreal corticosteroid injections) in the study eye OR participant has received any periocular or intravitreal injections in the fellow eye within the past 3 months
* Participant has evidence of previously active or currently active intraretinal neovascularization or subretinal neovascularization (SRNV), in either eye; subretinal or sub-RPE fibrovascular proliferation or disciform scars (subretinal fibrosis) in either eye are exclusionary;
* Participant has evidence of intraretinal hyperreflectivity** as evaluated by OCT in the study eye;
* Participant has a full thickness macular hole (FTMH) within the foveal area (ETDRS field 1) with a diameter of >400um at its narrowest point and outer retinal atrophy in the study eye;
* Amblyopia in the study eye; or
* Participant is allergic to fluorescein dye, and the clinical site does not have an OCT-A
* Participant has, in the opinion of the Investigator, any physical or mental condition that would increase the patient's risk of participation in the study or may interfere with the study procedures, evaluations and outcome assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
EZ loss | Baseline through Month 24
  Mean rate of change in the total area of EZ loss (IS/OS; macular photoreceptor loss) from Baseline (BL) through Month 24 (M24), as assessed using SD-OCT in the study eye(s).

SECONDARY OUTCOMES:
EZ loss at different time points | Baseline through Month 12 and 24
  Mean rate of change in the area of EZ loss (IS/OS; macular photoreceptor loss) from BL through Month 12 (M12) in the study eye(s) and through M12 and M24 in the fellow eye, as assessed using SD-OCT
Changes in Disease Severity | Baseline through Month 24
  Changes in disease severity (stages, according to Chew et al) in study eye(s), and fellow eye, from BL to M24
Retinal Sensitivity Loss | Baseline through Month 24
  Mean change in retinal sensitivity loss as measured by Macular Integrity Assessment (MAIA) from BL to M24 in study eye(s), and fellow eye
Reading Speed | Baseline through Month 24
  Mean change in monocular and binocular reading speed assessed using International Reading Speed Texts (IReST) cards from BL through M24 in the study eye(s), and fellow eye
Contrast Sensitivity | Baseline through Month 24
  Mean change in monocular contrast sensitivity from BL to M24 in the study eye(s) and fellow eye as assessed by Pelli-Robson contrast sensitivity charts
Low Luminance Visual Acuity | Baseline through Month 24
  Mean change in monocular low luminance visual acuity (LLVA) scores from BL to M24 in the study eye(s) and fellow eye as assessed by ETDRS charts
Low Luminance Deficit | Baseline through Month 24
  Mean change in low luminance deficit (LLVA - BCVA) from BL to M24 in the study eye(s) and fellow eye
Best Corrected Visual Acuity | Baseline through Month 24
  Mean change in monocular best-corrected visual acuity (BCVA) scores from BL to M24 in the study eye(s) and fellow eye as assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) charts
Corneal Nerve fiber Density | Baseline through Month 6, 12, 18 and 24
  Mean change in corneal nerve fiber and branch density (biomarkers of peripheral nerve health) from BL to M6, M12, M18 and M24 in the study eye(s) and fellow eye
HbA1c | Baseline through Months 12 and 24
  Mean change in HbA1c from BL to M12 and M24
BMI | Baseline through Months 12 and 24
  Mean change in BMI (weight and height will be combined to report BMI in kg/m^2) from BL to M12 and M24
Serum Metabolites | Baseline through Months 12 and 24
  Mean changes in fasted serum metabolite values from BL to M12 and M24
MacTel Metabolic Signature | Baseline through Months 12 and 24
  Mean changes in composite serum metabolic score measuring the global "MacTel Metabolic signature" from BL to M12 and M24
NEI VFQ-25 | Baseline through Month 12 and 24
  Mean change in NEI VFQ-25 scores from BL to M12 and M24
VILL-33 | Baseline through Months 12 and 24
  Mean change in VILL-33 scores from BL to M12 and M24
TEAEs and SAEs | Baseline through Month 24
  Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and ocular TEAEs and SAEs
ETDRS Letter Score | Baseline through Month 24
  Number of study eyes, fellow eyes with >= 15 letter loss (ETDRS letter score), >= 10 letter loss and >= 5 letter loss from BL to M24
Neovascularization | Baseline through Month 24
  Total number of study eyes, fellow eyes showing a de novo development of neovascularization from BL to M24
Outer Retinal Hyper-Reflectivity | Baseline through Month 24
  Total number of study eyes, fellow eyes showing a de novo development of outer retinal hyper-reflectivity from BL to M24
Hip to waist ratio | Baseline through Months 12 and 24
  Mean change in hip-to-waist ratio from BL to M12 and M24
Lipid Levels | Baseline through Months 12 and 24
  Mean change in Lipid Levels from BL to M12 and M24
Corneal Nerve Fiber Length | Baseline through Months 6, 12, 18 and 24
  Mean change in corneal nerve fiber length (biomarker of peripheral nerve health) from BL to M6, M12, M18 and M24 in the study eye(s) and fellow eye
Corneal Nerve Fiber Tortuosity | Baseline through Months 6, 12, 18 and 24
  Mean change in corneal nerve fiber tortuosity (biomarker of peripheral nerve health) from BL to M6, M12, M18 and M24 in the study eye(s) and fellow eye

CONTACTS AND LOCATIONS:
Locations (12):
- United States (4):
  - Hamilton Glaucoma Center- UCSD, La Jolla, California
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - Retina Associates Of Cleveland, Inc., Cleveland, Ohio
  - University of Utah Health Care, Moran Eye Center, Salt Lake City, Utah
- Australia (2):
  - Save Sight Institute, Sydney, New South Wales
  - Cerulea- RVEEH, Melbourne, Victoria
- Germany (3):
  - University of Bonn, Bonn
  - University of Freiburg, Department of Ophthalmology, Freiburg im Breisgau
  - St. Franziskus Hospital, Münster
- Radboud University Medical Center, Nijmegen, Netherlands
- United Kingdom (2):
  - Moorfields Eye Hospital, London
  - Oxford Eye Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No